CLINICAL TRIAL: NCT03531814
Title: Pilot Study of Medication Adherence in Children, Adolescents, and Adults With Neurofibromatosis Type 1 (NF1) on Clinical Treatment Trials
Brief Title: Medication Adherence in Children, Adolescents and Adults With Neurofibromatosis Type 1(NF1) on Clinical Treatment Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Staci Peron, Ph.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 180093; 18-C-0093
Record Dates: First submitted 2018-05-19; First posted 2018-05-22 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Neurofibromatosis 1; Neurofibroma, Plexiform
Keywords: Plexiform Neurofibromas; Medication Event Monitoring Systems; Oral Medication
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult Participants (Experimental): Questionnaires and use of the medication event monitoring system (MEMS^TM)
  Interventions: Behavioral: Medication Event Monitoring System (MEMS^TM); Other: Questionnaires
- Pediatric Participants 8+ Years (Experimental): Questionnaires and use of the medication event monitoring system (MEMS^TM)
  Interventions: Behavioral: Medication Event Monitoring System (MEMS^TM); Other: Questionnaires

INTERVENTIONS:
Behavioral: Medication Event Monitoring System (MEMS^TM) — A computerized method of tracking the dates and times of a pill bottle being opened.
Other: Questionnaires — Adult and pediatric participants completed a series of questionnaires to assess medication adherence, demographics, life events, and barriers to adherence.

SUMMARY:
Background:

Neurofibromatosis type 1 (NF1) is a genetic disorder. It has a broad variety of effects on the body. Up to half of people with NF1 get plexiform neurofibromas (PNs). These are benign tumors. But they can have serious effects like pain and disfigurement. To treat PNs, a person may have to take medicine every day for a long period of time. Researchers think that it will be important for people to take the medicine regularly for it to work. They want to study how well people with NF1 follow their treatment plan for PNs.

Objective:

To study how often people with neurofibromatosis type 1 take medicine that has been prescribed to them for treating plexiform neurofibromas.

Eligibility:

People ages 3-59 already enrolled in an NF1 clinical trial

Design:

Participants will need access to the internet to do the study activities.

Parents or caregivers will do some study activities for child participants.

Participants will complete 5 questionnaires. They will take about 20 minutes total. The topics will be:

Demographic data

Recent life events

How much pain interferes with daily life

Ability to focus and pay attention to tasks

Emotional distress or depression

Participants will mark down every time they take a dose of the medicine in their clinical trial. They will use a form the researchers give them. The pill bottles they get in their trial will have a chip in the cap that will record when it is opened. Participants will keep a daily diary of their medicine. Their pills will be counted at clinical trial visits.

Participants may have more short questionnaires. They may have interviews by phone or video.

DETAILED DESCRIPTION:
Background:

* Neurofibromatosis type 1 (NF1) is a genetic disorder that affects approximately 1 in 3,500 individuals and is associated with a broad variety of symptoms and physical findings.
* Plexiform neurofibromas (PN) are histologically benign tumors which occur in 25-50% of patients with NF1 and can lead to significant morbidity.
* Oral therapeutic options for the treatment of plexiform neurofibromas are being actively developed, however early clinical data indicate that prolonged treatment over the course of months to years will likely be needed to maintain clinical efficacy
* Long-term medication adherence is an ongoing challenge for patients with many types of chronic illness, and clinical experience makes us strongly suspect patients with NF1 will likely have this issue as well.
* In other diseases, such as human immunodeficiency virus (HIV) and Acute Lymphoblastic Leukemia, decreased medication adherence has been associated with poorer clinical outcomes, and this may be the case for NF1 as well.
* The medication event monitoring systems (MEMS^TM) uses a computerized method of tracking the dates and times of a pill bottle being opened and has been shown to be a more accurate measure of medication adherence than patient diaries or pill counts in other patient populations.
* Assessing medication adherence over time in this unique population will be essential for assessing any impact on medical outcomes, identifying potential behavioral interventions, and targeting patients most at risk for nonadherence moving forward.

Objective:

- To establish the feasibility of using MEMS^TM to monitor medication adherence in the NF1 population

Eligibility:

* Subjects must have a diagnosis of NF1 and be between 3 and 59 years of age
* Participants must be enrolled on a clinical trial for an oral medication in pill (tablet or capsule) form directed at the treatment of plexiform neurofibroma(s)

Design:

* This single-site, longitudinal study will recruit children and adults with NF1 who are currently enrolled in a treatment protocol for a drug targeting PN volume reduction.
* MEMS^TM caps will be used to monitor adherence over time along with patient diaries and pill counts.
* Patients with MEMS^TM cap data indicating <90% adherence at any study visit (typically across 3 - 6 cycles) will be administered a measure assessing barriers to adherence electronically and will be interviewed to evaluate what factors might contribute to decreased medication adherence and what potential interventions they consider useful.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Patient

* Patients must be between 3 and 59 years of age at the time of the baseline assessment.
* Patients must be enrolled on a neurofibromatosis Type 1 (NF1) clinical trial for an oral medication directed at the treatment of plexiform neurofibroma(s) (enrollment on this study to occur ideally within 1st cycle) Patients must have regular access to a computer or electronic device (e.g., smartphone, tablet) with internet access.
* Must have a parent or adult primary caregiver willing to participate in the study.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Subjects must be able to read and comprehend the English language.

Inclusion Criteria for Parents or Caregivers

* Must be a parent or primary caregiver of a child (or if applicable adult patient) of diagnosed with NF1 and enrolled on a clinical trial for oral medication.
* Must have a child (or if applicable adult patient) willing to participate in the study
* Must have regular access to a computer or electronic device (e.g., smartphone, tablet) with internet access.
* Must be able to speak and understand English.
* Ability of subject to understand and the willing to sign a written informed consent document.

EXCLUSION CRITERIA:

Exclusion Criteria for Patient

* In the opinion of the principal investigator (PI) or an associate investigator (AI), the subject has significant cognitive or emotional difficulties that would prevent them from being able to understand and/or participate fully in the study or complete the measures. Though these patients might be receiving assistance in taking medication from a caregiver, it is likely that their medication taking routine would be significantly different from the general population of patients with NF1.
* Patients receiving the study drug in liquid form, since the use of medication event monitoring systems (MEMS^TM) caps prohibits liquid dosing.

Exclusion Criteria for Parent or Caregiver

None

Ages: 3 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0093.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No pediatric participants were enrolled on this trial.
Groups:
- Adult Participants (18+ Years); Pediatric Participants (3-17 Years): Questionnaires and use of the medication event monitoring system (MEMS^TM)
  Participants must take an oral medication in pill (tablet or capsule) form directed at the treatment of plexiform neurofibroma(s).
  Medication Event Monitoring System (MEMS^TM) caps will be used to monitor adherence over time along with patient diaries and pill counts.
  Medication Event Monitoring System (MEMS^TM): A computerized method of tracking the dates and times of a pill bottle being opened.
Period: Overall Study
Arm/Group | Adult Participants (18+ Years) | Pediatric Participants (3-17 Years)
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.36 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Enrolled Participants for Which we Are Able to Collect Data From the Medication Event Monitoring Systems (MEMS^TM) System for Two or More Cycles of Treatment (Target = 75%)
Description: The proportion of enrolled participants are reported for individuals who had two full cycles of data recorded by the medication event monitoring systems (MEMS^TM) system. To monitor medication adherence the medication event monitoring system (MEMSTM) used to track the dates and times a pill bottle was opened. At least 2 cycles of medication adherence are considered a success.
Time Frame: Two cycles, approximately 56 days
Population: 11/12 participants were analyzed because 1 participant's cap malfunctioned, so no data was collected.
Measure: Number; unit: Proportion of participants
Groups:
- Adult Participants (18+ Years): Questionnaires and use of the medication event monitoring system (MEMS)
  Participants must take an oral medication in pill (tablet or capsule) form directed at the treatment of plexiform neurofibroma(s).
  Medication Event Monitoring System (MEMS) caps will be used to monitor adherence over time along with patient diaries and pill counts.
  Medication Event Monitoring System (MEMS): A computerized method of tracking the dates and times of a pill bottle being opened.
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Proportion of participants | 0.9167

2. Primary Outcome: Median Number of Cycles Monitored for Participants From the Medication Event Monitoring System (MEMS^TM)
Description: To monitor medication adherence the medication event monitoring system (MEMSTM) was used to track the dates and times a pill bottle was opened. We calculated the median number of cycles monitored for all patients.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: 11/12 participants were analyzed because 1 participant's cap malfunctioned, so no data was collected.
Measure: Median (Full Range); unit: Cycles
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Cycles | 16 [0 to 18]

3. Secondary Outcome: Average Percent Medication Adherence Over Time Based on the Medication Event Monitoring Systems (MEMS^TM) Pill Cap Data
Description: To monitor medication adherence the medication event monitoring system (MEMS^TM) was used to track the dates and times a pill bottle was opened. The number of times the bottle was opened was divided by the total number of times the bottle should be opened according to provider instructions. The mean of these numbers was computed across groups of cycles 1-4, 5-8, 9-12 and 13-18. A dose was considered adherent if it was taken within an 11-to-13-hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle and dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average. Higher number is better adherence.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: 11/12 participants (pts) analyzed Cycles(C) 1-4. 1 pts MEMS cap malfunctioned (= 0 data across any C). 10/12 pts analyzed C5-8. 1 additional pt withdrew from the study, resulting in 0 MEMS data beginning C5. 8/12 pts analyzed C9-12 & C13-18. 1 pt withdrew from study after C9 & 1 failed to return their MEMS Cap. Due to battery expiration between clinic visits, at least 1C was unable to be obtained for 5pts. And 1pt had missing data due to forgetting to replace the cap on the next cycle's bottle.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
percent
  Cycles 1-4 | 83.39 (16.71)
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 87.01 (14.62)
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | 84.77 (15.44)
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | 79.68 (20.85)

4. Secondary Outcome: ANOVA (Analysis of Variance) Comparing Average Adherence Measured by Medication Event Monitoring Systems (MEMS^TM), Medication Diary, and Pill Count
Description: A repeated-measures ANOVA was used to compare three adherence assessment methods over time. The medication event monitoring system (MEMS^TM) was used to track the dates and times a pill bottle was opened. The number of times the bottle was opened was divided by the total number of times the bottle should be opened according to provider instructions. Pill count was used to assess how many pills were returned at each restaging visit compared to the number that should be returned if all medication was taken as prescribed. The daily diary was completed by participants, documenting date and timing of doses. The mean of these numbers was computed across groups of cycles (1 cycle = 28 days) 1-4, 5-8, 9-12 and 13-18 for the MEMS^TM, Pill Count, and Daily Diary.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), an range of approximately 112 days to 504 days
Population: 11/12 participants (pts) analyzed Cycles(C) 1-4. 1 pts MEMS cap malfunctioned (= 0 data across any C). 10/12 pts analyzed C5-8 . 1 additional pt withdrew from the study, resulting in 0 MEMS data beginning C5. 8/12 pts analyzed C9-12 & C13-18. 1 pt withdrew from study after C9 & 1 failed to return their MEMS Cap. Due to battery expiration between clinic visits, at least 1C was unable to be obtained for 5pts. And 1pt had missing data due to forgetting to replace the cap on the next cycle's bottle.
Measure: Number; unit: ANOVA F-Value
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
ANOVA F-Value
  Cycles 1-4 | 11.944
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 7.770
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | 6.670
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | 6.333
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.006, ANOVA — The Greenhouse-Geisser correction was used because Mauchly's test of sphericity was significant. The reported p-value represents the probability of the differences in the averages of adherence assessment methods for cycles 1-4
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.021, ANOVA — The Greenhouse-Geisser correction was used because Mauchly's test of sphericity was significant. The reported p-value represents the probability of the differences in the averages of adherence assessment methods for cycles 5-8
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = .034, ANOVA — The Greenhouse-Geisser correction was used because Mauchly's test of sphericity was significant. The reported p-value represents the probability of the differences in the averages of adherence assessment methods for cycles 9-12
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = .040, ANOVA — The Greenhouse-Geisser correction was used because Mauchly's test of sphericity was significant. The reported p-value represents the probability of the differences in the averages of adherence assessment methods for cycles 13-18

5. Secondary Outcome: Spearman Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap and Age
Description: The outcome measures correlations between two variables and the resulting correlation coefficient describes the strength of the relationship between the variables. To assess the relationship between the adherence method MEMS^TM cap and age, Spearman correlation was used. For this analysis, MEMS^TM was defined as the average mean adherence for cycles 1-4, cycles 5-8, cycles 9-12, and cycles 13-18. A dose was considered adherent if it was taken within an 11-to-13-hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle and dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -0.210
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 0.134
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | .095
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | .333
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.536, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = -0.210, 95% CI 2-sided [-0.729 to 0.463]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = .713, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = 0.134, 95% CI 2-sided [-0.557 to 0.715]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = .823, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 9-12; Spearman's correlation = .095, 95% CI 2-sided [-0.668 to 0.761]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = .420, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = .333, 95% CI 2-sided [-0.505 to 0.848]

6. Secondary Outcome: Spearman Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap for Years of Education
Description: The outcome measures correlations between two variables and the resulting correlation coefficient describes the strength of the relationship between the variables. To assess the relationship between the adherence method MEMS^TM cap for years of education, Spearman correlation was used. For this analysis, MEMS^TM was defined as the average mean adherence for cycles 1-4. A dose was considered adherent if it was taken within an 11-to-13-hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle and dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average. Number of years of education was collected through participant self-report and was a continuous variable.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -0.333
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | -0.309
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | -0.259
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | -0.222
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.317, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = -0.333, 95% CI 2-sided [-0.785 to 0.352]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = .385, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = -0.309, 95% CI 2-sided [-0.794 to 0.416]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = .535, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 9-12; Spearman's correlation = -0.259, 95% CI 2-sided [-0.824 to 0.563]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = .597, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = -0.222, 95% CI 2-sided [-0.811 to 0.589]

7. Secondary Outcome: Spearman's Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap and Quality of Life (QOL) Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference T-scores
Description: Outcome measures correlations between 2 variables and the resulting correlation coefficient describes the strength of the relationship between the variables. To assess the relationship between the adherence method MEMS^TM cap & PROMIS Pain Interference T- Scores (Same for all PROMIS measures) Spearman correlation was used. For this analysis, MEMS^TM was defined as the average mean adherence for cycles 1-4. A dose was considered adherent if it was taken within an 11-13hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle & dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average. PROMIS Pain Interference raw scores transformed to T-scores for analysis (mean:50,standard deviation: 10, higher scores is more pain interference, T of 55 is cutoff-mild pain interference).
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -.215
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 0.049
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | -0.048
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | -0.167
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.526, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = -.215, 95% CI 2-sided [-0.731 to 0.459]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = .894, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = 0.049, 95% CI 2-sided [-0.613 to 0.670]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = .911, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 9-12; Spearman's correlation = -0.048, 95% CI 2-sided [-0.740 to 0.694]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = .693, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = -0.167, 95% CI 2-sided [-0.790 to 0.626]

8. Secondary Outcome: Spearman's Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap and Quality of Life (QOL) Patient-Reported Outcomes Measurement Information System (PROMIS) Depression T-scores
Description: The outcome measures correlations between two variables and the resulting correlation coefficient describes the strength of the relationship between the variables. To assess the relationship between the adherence method MEMS^TM cap and PROMIS Depression Scores, Spearman correlation was used. For this analysis, MEMS^TM was defined as the average mean adherence for cycles 1-4. A dose was considered adherent if it was taken within an 11-to-13-hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle and dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average. PROMIS Depression raw scores were transformed to T-scores for analysis (mean: 50, standard deviation: 10, higher scores is more depression symptoms, T of 55 is the cut off for mild depressive symptoms).
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficients
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficients
  Cycles 1-4 | -.607
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | -0.658
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | -0.708
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | -0.878
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.048, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = -.607, 95% CI 2-sided [-0.889 to 0.009]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.038, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = -0.658, 95% CI 2-sided [-0.914 to -0.027]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.50, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 9-12; Spearman's correlation = -0.708, 95% CI 2-sided [-0.945 to 0.020]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.004, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = -0.878, 95% CI 2-sided [-0.979 to -0.435]

9. Secondary Outcome: Spearman's Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap and Quality of Life (QOL) Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Interference T-scores
Description: The outcome measures correlations between two variables and the resulting correlation coefficient describes the strength of the relationship between the variables. To assess the relationship between the adherence method MEMS^TM cap and PROMIS Cognitive Interference Scores, Spearman correlation was used. For this analysis, MEMS^TM was defined as the average mean adherence for cycles 1-4. A dose was considered adherent if it was taken within an 11-to-13-hour interval from the prior correct dose. The mean was computed by summing medication adherence across the cycle and dividing it by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data to compute the average. PROMIS Cognitive Interference raw scores were transformed to T-scores for analysis (mean: 50, standard deviation: 10, higher scores is more cognitive interference, T of 60 represents mild interference).
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | 0.293
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 0.278
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | 0.229
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | 0.530
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.382, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = 0.293, 95% CI 2-sided [-0.390 to 0.768]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.436, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = 0.278, 95% CI 2-sided [-0.444 to 0.781]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.586, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 9-12; Spearman's correlation = 0.229, 95% CI 2-sided [-0.585 to 0.813]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.177, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = 0.530, 95% CI 2-sided [-0.302 to 0.904]

10. Secondary Outcome: Barriers to Adherence Questionnaire
Description: Participants completed a barriers questionnaire to assess barriers most frequently endorsed on the questionnaire. The questionnaire focused on any medication adherence issues during the trial (e.g., missed doses). Participants were given 16 possible reasons that they may have missed a dose and were asked to check all items that caused them to miss a dose of medication. Participants were also able to provide additional reasons for missing medication that were not on the form.
Time Frame: Baseline and follow-up (between cycles 8 and 12; or after cycle 18/when taken off of study (range of 224-504 days)
Population: Six participants were given the barriers to adherence questionnaire at baseline due to error. One participant was not given the barriers to adherence questionnaire at follow-up due to error, so only 11/12 participants had this at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Participants
  Most commonly reported barrier at baseline: Away from home: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Away from home | 0
  Most commonly reported barrier at baseline: Busy with other things: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Busy with other things | 0
  Most commonly reported barrier at baseline: Forgot: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Forgot | 0
  Most commonly reported barrier at baseline: Had too many pills to take: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Had too many pills to take | 0
  Most commonly reported barrier at baseline: Wanted to avoid having side effects: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Wanted to avoid having side effects | 0
  Most commonly reported barrier at baseline: Did not want others to see taking medication: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Did not want others to see taking medication | 0
  Most commonly reported barrier at baseline: Change in daily routine: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Change in daily routine | 0
  Most commonly reported barrier at baseline: Too tired or slept through dose time: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Too tired or slept through dose time | 0
  Most commonly reported barrier at baseline: Felt sick or ill: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Felt sick or ill | 0
  Most commonly reported barrier at baseline: Felt sad or stressed out: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Felt sad or stressed out | 0
  Most commonly reported barrier at baseline: Had problem taking medicine with clear liquid: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Had problem taking medicine with clear liquid | 0
  Most commonly reported barrier at baseline: Had difficulty swallowing pills: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Had difficulty swallowing pills | 0
  Most commonly reported barrier at baseline: Ran out of pills: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Ran out of pills | 0
  Most commonly reported barrier at baseline: Didn't like taste of medicine: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Didn't like taste of medicine | 0
  Didn't think medicine was working: number analyzed (Participants) | 6
  Didn't think medicine was working | 0
  Most commonly reported barrier at baseline: Didn't feel like it/Needed a break: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Didn't feel like it/Needed a break | 0
  Most commonly reported barrier at baseline: Other reason: number analyzed (Participants) | 6
  Most commonly reported barrier at baseline: Other reason | 0
  Most commonly reported barrier at follow-up: Forgetting | 6

11. Secondary Outcome: Spearman's Correlation of the Relationship Between Medication Event Monitoring Systems (MEMS^TM) Cap and Barriers to Adherence Questionnaire
Description: The outcome measures Spearman correlations between two variables and the resulting correlation coefficient describes the strength of the relationship between the variables. MEMS^TM was defined as the average mean adherence, an adherent dose was taken 11-13 hours from the prior correct dose. The mean was computed by dividing medication adherence across the cycle by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data. Barriers to adherence was calculated by summing the number of barriers for each participant at follow-up. Participants were given 16 possible reasons that they may have missed a dose and were asked to check all items that apply to them.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -0.576
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | -0.680
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | -0.835
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | -0.933
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.063, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 1-4; Spearman's correlation = -0.576, 95% CI 2-sided [-0.879 to 0.056]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.031, Wilcoxon (Mann-Whitney) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 5-8; Spearman's correlation = -0.680, 95% CI 2-sided [-0.920 to -0.066]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.010, Spearman correlation (non-parametric) — The reported p-value represents the strength of the relationship between the variables at cycles 9-12; Spearman's correlation = -0.835, 95% CI 2-sided [-0.971 to -0.292]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p < 0.001, Spearman correlation (non-parametric) — The reported p-value represents the probability that the strength of the relationship is due to chance at cycles 13-18; Spearman's correlation = -0.933, 95% CI 2-sided [-0.989 to -0.652]

12. Secondary Outcome: Medication Event Monitoring Systems (MEMS^TM) Cap and Stressful Life Events: Number of Stressful Life Events Endorsed in the Life Events Checklist
Description: To assess the relationship between the adherence method MEMS^TM cap and stressful life events (i.e., the number of stressful life events endorsed in the Life Events Checklist), Spearman correlation was used. Participants complete a 22-item questionnaire to report stressful events that impact medication adherence. MEMS^TM was defined as the average mean adherence, an adherent dose was taken 11-13 hours from the prior correct dose. The mean was computed by dividing medication adherence across the cycle by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -0.035
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | 0.227
  Cycles 9-12: number analyzed (Participants) | 8
  Cycles 9-12 | 0.179
  Cycles 13-18: number analyzed (Participants) | 8
  Cycles 13-18 | 0.041
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.919, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 1-4; Spearman's correlation = -0.035, 95% CI 2-sided [-0.634 to 0.591]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.528, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 5-8; Spearman's correlation = 0.227, 95% CI 2-sided [-0.487 to 0.759]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.672, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 9-12; Spearman's correlation = 0.179, 95% CI 2-sided [-0.618 to 0.794]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.923, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 13-18; Spearman's correlation = 0.041, 95% CI 2-sided [-0.697 to 0.737]

13. Secondary Outcome: Medication Event Monitoring Systems (MEMS^TM) Cap and Rating of Overall Stress
Description: To assess the relationship between the adherence method MEMS^TM cap and rating of overall stress, Spearman correlation was used. Participants complete a 1-item question asking them to rate their stress from 0 - 10, with higher numbers being more stressed. MEMS^TM was defined as the average mean adherence, an adherent dose was taken 11-13 hours from the prior correct dose. The mean was computed by dividing medication adherence across the cycle by the number of days within the cycle. Then, the average mean was calculated by using Statistical Package for the Social Sciences (SPSS) MEAN function, which uses all non-missing data.
Time Frame: Cycles 1-4, 5-8, 9-12 and 13-18 (1 cycle = 28 days), a range of approximately 112 days to 504 days
Population: as for outcome 4
Measure: Number; unit: Correlation coefficient
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 11
Correlation coefficient
  Cycles 1-4 | -0.638
  Cycles 5-8: number analyzed (Participants) | 10
  Cycles 5-8 | -0.361
  Cycles 9-12 | -0.407
  Cycles 13-18 | -0.180
Statistical Analysis 1: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.035, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 1-4; Spearman's correlation = -0.638, 95% CI 2-sided [-0.899 to -0.041]
Statistical Analysis 2: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.306, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 5-8; Spearman's correlation = -0.361, 95% CI 2-sided [-0.815 to 0.367]
Statistical Analysis 3: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.317, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 9-12; Spearman's correlation = -0.407, 95% CI 2-sided [-0.870 to 0.438]
Statistical Analysis 4: Comparison: Adult Participants (18+ Years); Test type: Other; p = 0.670, Spearman correlation — The reported p-value represents the strength of the relationship between the variables for cycles 13-18; Spearman's correlation = -0.180, 95% CI 2-sided [-0.795 to 0.0617]

14. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events
Description: Here is the number of participants with serious and/or non-serious adverse events. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Baseline to cycle 18 (end of study), approximately 504 days (1.38 years)
Population: As pre-specified by the protocol, adverse events occurring because of treatment for the underlying condition or medical treatment for pain will NOT be recorded in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants (18+ Years)
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline to cycle 18 (end of study), approximately 504 days (1.38 years)
Description: As pre-specified by the protocol, adverse events occurring as a result of treatment for the underlying condition or medical treatment for pain will NOT be recorded on this study.
Arm/Group | Adult Participants (18+ Years)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03531814/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT03531814/ICF_001.pdf